CLINICAL TRIAL: NCT04754139
Title: A Promotion and Implementation Project of HIV Pre-Exposure Prophylaxis Among High Risk Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Gilead Sciences (Industry); Guangzhou 8th People's Hospital (Other); Social Entrepreneurship to Spur Health (Other); Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB20-1388
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: HIV Preexposure Prophylaxis
Keywords: Preexposure prophylaxis (PrEP), Prevention, mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeChat mobile mini-application (Experimental): WeChat mini-application will increase knowledge base about sexual health through interactive health education and counseling support on HIV/STI prevention as well as PrEP initiation and/or adherence management.
  Interventions: Other: WeChat mobile mini-application

INTERVENTIONS:
Other: WeChat mobile mini-application — Sexual health education and the role of PrEP

SUMMARY:
This study aims to use a social media mini-application-enabled intervention to successfully promote the initiation and persistence of pre-exposure prophylaxis (PrEP) among at-risk people 18 years and above (including men who have sex with men (MSM), transgender women, sex workers, and other key populations) in Wuhan and Guangzhou, China.

DETAILED DESCRIPTION:
The China National Medical Products Administration (NMPA) recently approved TDF/FTC (Truvada) for PrEP making it the first HIV prevention medicine available in China. While this is a significant step in addressing the country's rising rates of new HIV diagnoses, implementation and scale-up of this resource will be the next challenge.

3200 at-risk adults will be engaged by word of mouth and social media. Individuals will be asked to complete a survey of risk and PrEP interest, to download the study mobile mini-application onto their cell phone, and will be offered an HIV and syphilis screen. One thousand two hundred of these subjects who are eligible and willing to start PrEP will be enrolled in the study. The first 700 participants enrolled in each site will complete an additional four-phased, WeChat-based adherence intervention through a stepped-wedge design, with each cluster starting at three-month intervals.

Enrolled participants will undergo baseline laboratory testing before brought to a collaborating hospital where an established physician will provide TDF/FTC and arrange follow-up. Rural and out-of-town enrollees may undergo testing at an outside lab. All subjects will be encouraged to keep using the mini-application for receiving constant health education and counseling support on HIV/STI prevention, PrEP initiation and/or adherence management. Subjects on PrEP will be contacted every three months over the course of two years to answer questions on adherence including number of missed pills and/or sex events not covered by on-demand PrEP, adverse effect, and utilization of the mini-application. 120 enrollees in Guangdong will additionally participate in a pill count adherence sub study that counts the number of unused pills at each clinical follow-up

A PrEP messaging open contest will be organized to assess the best images and videos to enhance PrEP adherence among those who start PrEP. New content will be developed using crowdsourcing and introduced into the mini-application at staggered times. The effect of this content will be evaluated through a stepped wedge approach nested within this single arm study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Engaged in at-risk sex. At risk sex is defined as sex with >1 partner in the past 90 days, inconsistent condom use with vaginal or anal sex, ongoing sexual relationship with an HIV-positive partner, participation in commercial sex work, or any bacterial STI diagnosed or reported in the past 6 months.

Exclusion Criteria:

* History renal dysfunction
* Chronic hepatitis B (HBV) infection
* HIV infection
* Indication for HIV post-exposure prophylaxis
* Signs and symptoms consistent with acute HIV infection
* Under the age range of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
PrEP prescriptions | 2 years
  Number of PrEP prescriptions fulfilled in Wuhan and Guangzhou, China

SECONDARY OUTCOMES:
HIV Screenings | 2 years
  Number of HIV screenings performed
Syphilis screenings | 2 years
  Number of syphilis screenings performed
Retention | 12 months
  Number of subjects retained in PrEP care at 6 and 12 months
Adherence | 2 years
  Number of subjects that self-report PrEP adherence
New HIV infection | 2 years
  Number of new HIV infections reported in PrEP users
New syphilis infection | 2 years
  Number of new syphilis infections reported in PrEP users

CONTACTS AND LOCATIONS:
Overall Officials: Aniruddha Hazra, MD, Principal Investigator — University of Chicago
Locations (2):
- China (2):
  - Guangzhou Eighth People's Hospital, Guangzhou
  - Zhongnan Hospital of Wuhan University, Wuhan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sha Y, Li C, Xiong Y, Hazra A, Lio J, Jiang I, Huang H, Kerman J, Molina J, Li L, Liang K, Gong D, Li Q, Wu S, Sherer R, Tucker JD, Tang W. Co-creation using crowdsourcing to promote PrEP adherence in China: study protocol for a stepped-wedge randomized controlled trial. BMC Public Health. 2022 Sep 7;22(1):1697. doi: 10.1186/s12889-022-14117-5. PMID 36071401